CLINICAL TRIAL: NCT05217901
Title: A Phase 1, Open-label Study to Evaluate the Absorption, Metabolism and Excretion of [14C]ASP0367 Solution in Healthy Male Participants
Brief Title: A Study to Learn How [14C]ASP0367 is Processed by the Body in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0367-CL-1103
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Healthy Volunteers; ASP0367; MA-0211

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 14C-labeled ASP0367 (Experimental): Participants will receive a single oral dose of [14C]ASP0367 solution under fasting conditions on day 1.
  Interventions: Drug: 14C-labeled ASP0367

INTERVENTIONS:
Drug: 14C-labeled ASP0367 — Oral
  Other Names: MA-0211; bocidelpar

SUMMARY:
ASP0367 is a potential new treatment for people with Duchenne Muscular Dystrophy and Mitochondrial Myopathies. Before ASP0367 is available as a treatment, the researchers need to understand how it is processed by and acts upon the body. This study is in healthy men.

The main aim of this study is to learn how ASP0367 is processed by and acts upon the bodies of healthy men. To do this, [14C] which is a certain chemical (called a tracer, or radionuclide) has been added to ASP0367. [14C] gives off radiation, but the dose is very low (about the same as the dose from an x-ray) and will leave the body within a few days. [14C] will be picked up by a scanner and will be used to follow ASP0367 through the body. [14C]ASP0367 will be a liquid.

During the study, the men who take part will stay in the clinic for 6 days and 5 nights. Some men may need to stay up to an extra 7 days in the clinic. This will happen if there is a medical reason or if they still have traces of radiation in their blood, urine or feces. On the day before they drink [14C]ASP0367, the men will be asked about their medical history, have a medical examination, and have their vital signs checked (blood pressure and pulse). They will also have an ECG to check their heart rhythm. They will give urine, stool and blood samples for laboratory tests. They will also be asked if they have had any medical problems.

The men will fast for 10 hours or more before drinking [14C]ASP0367 and for 4 hours afterwards. They will only have one drink of [14C]ASP0367. They will need to lie still for 4 hours after drinking [14C]ASP0367. They will have their vital signs checked and give urine, stool and blood samples for laboratory tests. Then, they will give urine, stool and blood samples every day until they leave the clinic. They will also be asked every day if they have had any medical problems.

The day after they drink [14C]ASP0367, the men will also have an ECG. On the last clinic day, the men will also have a physical exam, have their vital signs checked and have an ECG. The men can leave the clinic once [14C]ASP0367 has left the body and they have no medical problems.

About 10 days later, the clinic will call the men to check if there were any further medical problems.

No other visits are planned during this study.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a body mass index range of 18.5 to 32.0 kg/m^2 inclusive and weighs at least 50 kg at screening.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner[s]) must agree to use contraception throughout the treatment period and for 90 days after investigational product (IP) administration.
* Male participant must not donate sperm during the treatment period and for 90 days after IP administration.
* Male participant with pregnant partner(s) must agree to use a condom and spermicide for the duration of the pregnancy throughout the study and for 90 days after IP administration.
* Participant has regular bowel habits (i.e., at least 1 bowel movement per day).
* Participant agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Participant has received any investigational therapy within 28 days or 5 half lives, whichever is longer, prior to screening.
* Participant has participated in more than 3 radiolabeled studies within 12 months prior to day -1 (participation in a previous radiolabeled study has to have been at least 4 months prior to day -1 where exposures are known to the investigator, or 6 months prior to day -1 where exposures are not known to the investigator). The cumulative annual radiation exposure from this study and a maximum of 3 previous radiolabeled studies within 12 months prior to day -1 will be within the recommended level of radiation exposure considered to be safe.
* Participant has exposure to significant diagnostic or therapeutic radiation (e.g., serial X ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to day -1.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to ASP0367 or any components of the formulation used.
* Participant has had previous exposure with ASP0367.
* Participant has any of the liver function tests (alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase and total bilirubin) ≥ 1.5 x upper limit of normal (ULN) on day -1. In such a case, the assessment may be repeated once.
* Participant has creatinine level outside normal limits on day -1. In such a case, the assessment may be repeated once.
* Participant has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to IP administration.
* Participant has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Participant has any history or evidence of Gilbert's Disease.
* Participant has previously undergone a cholecystectomy.
* Participant has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to day -1.
* Participant has any clinically significant abnormality following the physical examination on day -1 and electrocardiogram (ECG) and protocol defined clinical laboratory tests at screening or on day -1.
* Participant has a mean pulse < 45 or > 90 bpm; mean systolic blood pressure > 140 mmHg; mean diastolic blood pressure > 90 mmHg (measurements taken in triplicate after participant has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional triplicate may be taken.
* Participant has a mean corrected QT interval using Fridericia's formula (QTcF) of > 430 msec on day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG may be taken.
* Participant has used any prescribed or nonprescribed drugs (including vitamins and natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to IP administration, except for occasional use of acetaminophen (up to 2 g/day), topical dermatological products (including corticosteroid products).
* Participant has smoked, used tobacco containing products and nicotine or nicotine containing products (e.g., electronic vapes) within 6 months prior to screening or the participant tests positive for cotinine at screening or on day -1.
* Participant has a history of consuming > 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within 2 years prior to screening (note: 1 unit = 12 ounces of beer, 4 ounces of wine, 1 ounce of spirits/hard liquor) or the participant tests positive for alcohol at screening or on day -1.
* Participant has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) within 3 months prior to day -1 or the participant tests positive for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and/or opiates) at screening or on day -1.
* Participant has used any inducer of metabolism (e.g., barbiturates and rifampin) in the 3 months prior to day -1.
* Participant has had significant blood loss, donated ≥ 1 unit (450 mL) of whole blood or donated plasma within 7 days prior to day -1 and/or received a transfusion of any blood or blood products within 60 days.
* Participant has a positive serology test for hepatitis A virus antibodies immunoglobulin M, hepatitis B core antibodies, hepatitis B surface antigen, hepatitis C virus antibodies or antibodies to human immunodeficiency virus type 1 and/or type 2 at screening.
* Participant is an employee of Astellas, the study-related contract research organizations or the clinical unit.
* Participant has consumed grapefruit/Seville orange or grapefruit/Seville orange containing products within 72 hours prior to day -1.
* Participant has received a coronavirus disease 2019 (COVID 19) vaccine within the 2 weeks prior to IP administration or will have a COVID 19 vaccine dose before the end of study telephone call.
* Participant has a positive result for severe acute respiratory syndrome coronavirus 2 test at screening or on day -1.
* Participant has cardiac troponin I (cTnI) > ULN [or cardiac troponin T > ULN if cTnI is not available] at screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of 14C-labeled ASP0367 (radioactivity in whole blood): Area Under The Concentration Time curve From The Time of Dosing Extrapolated to Time Infinity (AUCinf) | Up to 12 days
  AUCinf will be recorded from PK whole blood samples collected.
PK of 14C-labeled ASP0367 (radioactivity in whole blood): Area Under The Concentration-time Curve From The Time of Dosing to The Last Measurable Concentration (AUClast) | Up to 12 days
  AUClast will be recorded from PK whole blood samples collected.
PK of 14C-labeled ASP0367 (radioactivity in whole blood): Maximum Concentration (Cmax) | Up to 12 days
  Cmax will be recorded from PK whole blood samples collected.
Pharmacokinetics (PK) of 14C-labeled ASP0367 (radioactivity in plasma): AUCinf | Up to 12 days
  AUCinf will be recorded from PK plasma samples collected.
Pharmacokinetics (PK) of 14C-labeled ASP0367 (radioactivity in plasma): AUClast | Up to 12 days
  AUCinf will be recorded from PK plasma samples collected.
Pharmacokinetics (PK) of 14C-labeled ASP0367 (radioactivity in plasma): Cmax | Up to 12 days
  AUCinf will be recorded from PK plasma samples collected.
PK of 14C-labeled ASP0367 (radioactivity ratio of whole blood/plasma concentrations) in blood: Radioactivity Ratio of Area Under The Concentration Time Curve in Blood as Compared to Plasma (AUCblood/AUCplasma) | Up to 12 days
  AUCblood/AUCplasma will be recorded from PK whole blood and plasma samples collected.
Excretion of 14C-labeled ASP0367 (radioactivity in urine): amount of administered dose excreted (Ae) | Up to 12 days
  Ae will be recorded from urine samples collected.
Excretion of 14C-labeled ASP0367 (radioactivity in urine): percentage of administered dose excreted (Ae percentage) | Up to 12 days
  Ae percentage will be recorded from urine samples collected.
Excretion of 14C-labeled ASP0367 (radioactivity in urine): cumulative (over more than 1 sampling interval) amount of administered dose excreted (CumAe) | Up to 12 days
  CumAe will be recorded from urine samples collected.
Excretion of 14C-labeled ASP0367 (radioactivity in urine): cumulative (over more than 1 sampling interval) percentage of administered dose excreted (CumAe percentage) | Up to 12 days
  CumAe percentage will be recorded from urine samples collected.
Excretion of 14C-labeled ASP0367 (radioactivity in urine): renal clearance (CLR) | Up to 12 days
  CLR will be recorded from urine samples collected.
Excretion of 14C-labeled ASP0367 (radioactivity in feces): Ae | Up to 12 days
  Ae will be recorded from feces samples collected.
Excretion of 14C-labeled ASP0367 (radioactivity in feces): Ae percentage | Up to 12 days
  Ae percentage will be recorded from feces samples collected.
Excretion of 14C-labeled ASP0367 (radioactivity in feces): CumAe | Up to 12 days
  CumAe will be recorded from feces samples collected.
Excretion of 14C-labeled ASP0367 (radioactivity in feces): CumAe percentage | Up to 12 days
  CumAe percentage will be recorded from feces samples collected.
Excretion of 14C-labeled ASP0367 (radioactivity in emesis): Ae | Up to 12 days
  Ae (if applicable) will be recorded from emesis samples collected.
Excretion of 14C-labeled ASP0367 (radioactivity in emesis): Ae percentage | Up to 12 days
  Ae percentage (if applicable) will be recorded from emesis samples collected.
Excretion of 14C-labeled ASP0367 (radioactivity in emesis): CumAe | Up to 12 days
  CumAe (if applicable) will be recorded from emesis samples collected.
Excretion of 14C-labeled ASP0367 (radioactivity in emesis): CumAe percentage | Up to 12 days
  CumAe percentage(if applicable) will be recorded from emesis samples collected.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 23 days
  An AE will be coded using MedDRA. An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of IP, whether or not considered related to the IP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP. This includes events related to the comparator and events related to the (study) procedures.
Number of Participants with Laboratory Value Abnormalities and/or AEs | Up to 12 days
  Number of participants with potentially clinically significant laboratory values.
Number of Participants with Vital Sign Abnormalities and/or AEs | Up to 5 days
  Number of participants with potentially clinically significant vital sign values.
Number of Participants with 12-Lead Electrocardiogram (ECG) Abnormalities and/or AEs | Up to 5 days
  Number of participants with potentially clinically significant 12-Lead ECG values.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Labcorp CRU, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.